CLINICAL TRIAL: NCT04846166
Title: Role of Inhibitor SMADs in Stage 3 Grade B Periodontitis Before and After Periodontal Treatment
Brief Title: I-Smads in Periodontitis
Status: Completed | Type: Observational
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Figen Öngöz Dede, T.C. ORDU ÜNİVERSİTESİ, Bulent Ecevit University
Other Study IDs: B-1921
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Periodontitis; Treatment Adherence
Keywords: Smad; Periodontitis; Gingival crevicular fluid; Saliva
MeSH Terms: conditions — Periodontitis; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control
  Interventions: Diagnostic Test: Periodontally healthy group
- Periodontitis
  Interventions: Diagnostic Test: Periodontitis

INTERVENTIONS:
Diagnostic Test: Periodontally healthy group — probing pocket depth (PPD)≤ 3 mm (presence of normal gingival sulcus), bleeding on probing (BOP) < 10%, clinical absence of periodontal inflammation, radiological bone loss, and any prior periodontal disease, additionally presence of anatomically intact periodontium
  Groups: Control
Diagnostic Test: Periodontitis — : interdental clinical attachment level (CAL) ≥ 5 mm and PPD ≥ 6 mm on at least two non-adjacent teeth, bone loss involving the middle or apical third of the root radiographically, moderate ridge defect and ≥30% of teeth
  Groups: Periodontitis

SUMMARY:
Recently, it has been stated that Smads play an active role in all conditions where transforming growth factor-beta (TGF-β) is involved, including periodontal inflammation. This study aimed to examine the levels of TGF-β and inhibitor Smads in saliva and gingival crevicular fluid (GCF) in patients with Stage 3 Grade B periodontitis before and after non-surgical periodontal treatment. Twenty (20) stage 3 grade B periodontitis and 20 periodontally healthy individuals were included in the study. Clinical periodontal measurements were recorded; periodontitis patients received non-surgical periodontal treatment, and GCF and saliva samples were obtained at baseline and one month after treatment. TGF-β, Smad6, and Smad7 were determined by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Have at least 20 natural teeth, excluding third molars.
* Periodontitis patients had at least two non-adjacent sites per quadrant with probing depth (PD) ≥ 5 mm and clinical attachment level (CAL) ≥ 5 mm with gingival inflammation, and alveolar bone loss affecting >30% of the teeth, as detected on clinical and radiographical examinations.
* Periodontally healthy control group had no sign of gingival inflammation, no PD > 3mm and no evidence of attachment or bone loss

Exclusion Criteria:

* History of systemic disease.
* Regular use of any drugs which can effect the immune system or inflammatory response in the 6 months preceding the start of the study.
* Periodontal treatment during last 6 months that could affect periodontal status.
* Smoking.
* History of radiotherapy or chemotherapy.
* Current pregnancy, lactation or menopause.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. group (Control): Periodontally and systemically healthy
  2. group: Systemically healthy and periodontitis
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
TGF-β, Smad6, and Smad7 levels | baseline
  the levels of TGF-β, Smad6, and Smad7 in gingival crevicular fluid (GCF) and saliva

SECONDARY OUTCOMES:
TGF-β, Smad6, and Smad7 levels | baseline and 1st month after treatment
  the levels of TGF-β, Smad6, and Smad7 in gingival crevicular fluid (GCF) and saliva before and after non-surgical periodontal treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Figen Öngöz Dede, Ordu, Turkey (Türkiye)